CLINICAL TRIAL: NCT05038163
Title: Are Sugar-Sweetened Beverage Information Labels Well-Targeted: Evidence and Welfare Implications
Brief Title: Are Sugar-Sweetened Beverage Information Labels Well-Targeted
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: University of California, Berkeley (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-08-13558; P30AG034532 (NIH)
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Soft Drink Consumption; Sugar-sweetened Beverages; Information Labels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Arm (No Intervention): In Part II of the experiment, subjects are not presented with nutrition or warning labels when choosing between beverages.
- Nutrition Labels Arm (Experimental): In Part II of the experiment, subjects are shown enlarged nutrition labels when choosing between beverages.
  Interventions: Other: Nutrition Facts
- Text Warning Labels Arm (Experimental): In Part II of the experiment, subjects are shown a warning message about the health risks of sugary beverages when choosing between beverages.
  Interventions: Other: Text Warning
- Graphic Warning Labels Arm (Experimental): In Part II of the experiment, subjects are shown a graphic warning message about the health risks of sugary beverages when choosing between beverages. The message, for example, could include photos of tooth decay and other negative health outcomes.
  Interventions: Other: Graphic Warning

INTERVENTIONS:
Other: Nutrition Facts — The nutritional information label for each beverage is enlarged.
  Arms: Nutrition Labels Arm
Other: Text Warning — The health risks of sugary beverages are communicated to subjects using words/text and simple images.
  Other Names: Stoplight Warning
  Arms: Text Warning Labels Arm
Other: Graphic Warning — The health risks of sugary beverages are communicated to subjects using a combination of words/text and graphic images/photographs.
  Arms: Graphic Warning Labels Arm

SUMMARY:
We will study the extent to which soft drink information labels -- designed to curb unhealthy consumption -- are well-targeted to the most biased consumers.The study team will deploy novel methods for evaluating the targeting properties of information labels via an incentive-compatible online shopping experiment. At a high-level, we will ask whether the treatment effects of the information labels are concentrated on individuals with the biggest self-control problems and with the least knowledge of nutrition. We will first use the methodology from Allcott et al. (2019) to estimate the internality for each participant. We will then have participants make shopping decisions for soft drinks, first absent any information labels and then, for those not in the control group, in the presence of an information label. The within-subject design of the soft drinks experiment will allow us to estimate how the effects of the labels covary with consumers' internalities, and thus to determine whether the labels are well-targeted.

DETAILED DESCRIPTION:
We will use online ads to recruit people who are shopping online for soda, and direct them to a two-stage online Qualtrics experiment. In the first stage (Part I), we will elicit subjects' nutritional literacy and self-control for resisting sugary drinks, following the methodology of Allcott et al. (2019). Allcott et al. (2019) show that these two measures explain 31% of sugary drinks consumption in a nationally-representative sample of approximately 20,000 households, after controlling for detailed demographic information and elicitations of "tastes" for various types of drinks. Additionally, Allcott et al. (2019) demonstrate how these measures can be used to provide an estimate of over-consumption of sugary drinks at the individual level. Consequently, the first stage allows us to obtain estimates of the internality.

A week later, we will recruit participants in the first stage to participate in the second stage of the experiment (Part II). We create a time delay to minimize the potential effect of the first-stage questions on the second-stage choices. In the second stage, we will first ask participants to select their three favorite sugary drinks from a list. We will then ask participants to make an initial set of choices between those drinks and sugar-free alternatives (e.g., Seagram's Ginger Ale versus 365 Ginger) at various relative prices. Specifically, we will elicit their willingness to pay using a multiple price list, as is standard in the behavioral economics literature, where consumers answer a series of questions about whether they would prefer to buy a sugar-sweetened beverage at price X or a sugar-free alternative at price Y. Choices will be incentive-compatible: for each consumer we will honor their choice in a randomly selected decision (i.e., we will purchase the chosen package of soft drinks for them plus award them any additional money associated with that choice).

Following an initial set of choices, we will ask subjects to choose again. In this second set of choices, we will randomize whether participants see the soft drink options paired with an information label. We will also randomize the types of labels, including: (i) an inflated nutrition label that draws attention to the differences in calories and sugar content, (ii) the stoplight warning label developed by Grummon, Hall, et al. (2019), and (iii) a graphic warning label developed by Donnelly et al. (2018). The control group will instead make the same choices without seeing any label. Leveraging the within-subject nature of design, we will then estimate how well-targeted each information label is by estimating how the subjects' internalities covary with their changes in the prices at which they are willing to buy soft drinks after seeing the information label.

ELIGIBILITY:
Inclusion Criteria:

* US resident
* Shopping online for sugar-sweetened beverages

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5845 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Taubinsky, PhD, Principal Investigator — UC Berkeley and NBER
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be posted to ClinicalTrials.gov and Open Science Framework within 12 months of the primary completion date or the resulting paper's online publication date, whichever comes first.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 12 months of the primary completion date or the resulting paper's online publication date, whichever comes first.
Access Criteria: Replication data and code are available via Dropbox. Use the URL provided below, or navigate to the project by searching for "When Do 'Nudges' Increase Welfare?" at allcott.stanford.edu/research/.
URL: https://www.dropbox.com/scl/fi/t6flwxjy57ek74dxtvom7/OptimalNPI_replication.zip?rlkey=j564xs9k6ftwi64fll417aroh&e=1&dl=0

REFERENCES:
- [Background] Allcott H, Lockwood BB, Taubinsky D. Regressive Sin Taxes, with an Application to the Optimal Soda Tax. Quarterly Journal of Economics. 2019; 134(3).
- [Background] Grummon AH, Hall MG, Taillie LS, Brewer NT. How should sugar-sweetened beverage health warnings be designed? A randomized experiment. Prev Med. 2019 Apr;121:158-166. doi: 10.1016/j.ypmed.2019.02.010. Epub 2019 Feb 14. PMID 30772370
- [Background] Donnelly GE, Zatz LY, Svirsky D, John LK. The Effect of Graphic Warnings on Sugary-Drink Purchasing. Psychol Sci. 2018 Aug;29(8):1321-1333. doi: 10.1177/0956797618766361. Epub 2018 Jun 18. PMID 29912624

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a two-stage study. In Stage 1, participants completed a baseline survey about their demographic characteristics, consumer bias, self control, and nutrition knowledge. Randomization occurred in Stage 2, in which participants' willingness to pay for sugary drink was measured.
Groups:
- Stage 1 - All Enrolled Participants: Baseline survey about demographic characteristics, consumer bias, self control, and nutrition knowledge
- Stage 2 - Not Randomized: Subjects began Part II of the experiment, but did not reach the point of randomization.
Period: Stage 1
Arm/Group | Stage 1 - All Enrolled Participants | Control Arm | Graphic Warning Labels Arm | Nutrition Labels Arm | Text Warning Labels Arm | Stage 2 - Not Randomized
Started | 4033 | 0 | 0 | 0 | 0 | 0
Completed | 3659 | 0 | 0 | 0 | 0 | 0
Not Completed | 374 | 0 | 0 | 0 | 0 | 0
Not completed — Did not complete survey | 374 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1 - All Enrolled Participants | Control Arm | Graphic Warning Labels Arm | Nutrition Labels Arm | Text Warning Labels Arm | Stage 2 - Not Randomized
Started | 0 | 696 | 683 | 668 | 683 | 100
Completed | 0 | 667 | 653 | 644 | 662 | 0
Not Completed | 0 | 29 | 30 | 24 | 21 | 100
Not completed — Did not complete Stage 2 survey | 0 | 29 | 30 | 24 | 21 | 100

BASELINE CHARACTERISTICS:
Population: Includes all participations who completed the Stage 1 survey.
Groups:
- Non-Randomized: Subjects did not reach Part II and were therefore not randomized.
- Total: Total of all reporting groups
Arm/Group | Control Arm | Graphic Warning Labels Arm | Nutrition Labels Arm | Text Warning Labels Arm | Non-Randomized | Total
Number analyzed (Participants) | 667 | 653 | 644 | 662 | 1033 | 3659
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 3 | 4 | 2 | 18
  Between 18 and 65 years | 535 | 527 | 526 | 551 | 680 | 2819
  >=65 years | 129 | 120 | 115 | 107 | 351 | 822
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.97 (16.60) | 48.39 (16.71) | 49.04 (16.80) | 47.48 (16.52) | 58.49 (14.17) | 51.12 (16.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Includes respondents who answered Female or Male to question about gender
  Participants
    number analyzed (Participants) | 655 | 637 | 631 | 652 | 1023 | 3598
    Female | 339 | 323 | 327 | 354 | 602 | 1945
    Male | 316 | 314 | 304 | 298 | 421 | 1653
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 26 | 27 | 48 | 37 | 166
  Not Hispanic or Latino | 601 | 592 | 584 | 595 | 873 | 3245
  Unknown or Not Reported | 38 | 35 | 33 | 19 | 123 | 248
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 6 | 5 | 5 | 15 | 40
  Asian | 34 | 37 | 37 | 40 | 24 | 172
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 1 | 3 | 8
  Black or African American | 17 | 29 | 24 | 25 | 32 | 127
  White | 563 | 551 | 548 | 551 | 899 | 3112
  More than one race | 26 | 18 | 14 | 19 | 30 | 107
  Unknown or Not Reported | 17 | 11 | 14 | 21 | 30 | 93
Bias [Mean (Standard Deviation); unit: Dollars per 12-pack of soda] — Survey-based estimate of consumer bias, the amount by which consumers over-estimate their utility from consuming sugary drinks
  Dollars per 12-pack of soda | 2.60 (1.24) | 2.52 (1.22) | 2.52 (1.28) | 2.58 (1.22) | 2.70 (1.28) | 2.56 (1.24)
Self-Control [Mean (Standard Deviation); unit: units on a scale] — Survey-based estimate of self-control. Participants were asked to respond to the statement "I drink soda pop or other sugar-sweetened beverages more often than I should," with possible responses of "Definitely," "Mostly," "Somewhat," and "Not at all." These answers were coded as 0, 1/3, 2/3, and 1, respectively.
  units on a scale | 0.40 (0.37) | 0.41 (0.37) | 0.41 (0.37) | 0.40 (0.36) | 0.39 (0.37) | 0.41 (0.37)
Nutrition Knowledge [Mean (Standard Deviation); unit: Proportion of correct answers] — Participants were asked to answer 28 questions from the General Nutrition Knowledge Questionnaire (GNKQ), a widely used nutrition-knowledge elicitation device in the public health literature. Each participant's nutrition knowledge score was then estimated as the proportion of correct answers among the 28. Hence higher values represent greater nutrition knowledge.
  Proportion of correct answers | 0.69 (0.12) | 0.70 (0.11) | 0.70 (0.12) | 0.69 (0.12) | 0.67 (0.12) | 0.68 (0.14)

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Purchase Sugar-sweetened Beverage vs. Sugar-free Alternative
Description: How much consumers like, or are willing to pay for, sugar-sweetened beverages when compared to a sugar-free alternative. The survey instrument uses a multiple price list (MPL) to elicit each respondent's relative willingness to pay (WTP) for the sugary drink vs. the non-sugary alternative, a standard methodology in the economics literature where consumers answer a series of questions about whether they would prefer to buy a sugar-sweetened beverage at price X or a sugar-free alternative at price Y. For example, a relative WTP of $1.60 indicates a respondent is willing to pay an additional $1.60 for the sugary drink compared to the non-sugary alternative.
Time Frame: 1 week after recruitment (during Part II of the experiment)
Measure: Mean (Standard Deviation); unit: Dollars per 12-pack of soda
Arm/Group | Control Arm | Graphic Warning Labels Arm | Nutrition Labels Arm | Text Warning Labels Arm
Number analyzed (Participants) | 667 | 653 | 644 | 662
Dollars per 12-pack of soda | 0.06 (0.84) | -0.46 (1.34) | -0.39 (1.23) | -0.29 (1.03)
Statistical Analysis 1: Comparison: Control Arm vs Graphic Warning Labels Arm; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.51, 95% CI 2-sided [-0.63 to -0.39]
Statistical Analysis 2: Comparison: Control Arm vs Nutrition Labels Arm; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.45, 95% CI 2-sided [-0.57 to -0.33]
Statistical Analysis 3: Comparison: Control Arm vs Text Warning Labels Arm; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.34, 95% CI 2-sided [-0.44 to -0.24]

2. Primary Outcome: Willingness to Purchase Sugar-sweetened Beverage vs. Sugar-free Alternative, Among Adults Aged 65+
Description: How much older adult consumers like, or are willing to pay for, sugar-sweetened beverages when compared to a sugar-free alternative. The survey instrument uses a multiple price list (MPL) to elicit each respondent's relative willingness to pay (WTP) for the sugary drink vs. the non-sugary alternative, a standard methodology in the economics literature where consumers answer a series of questions about whether they would prefer to buy a sugar-sweetened beverage at price X or a sugar-free alternative at price Y. For example, a relative WTP of $1.60 indicates a respondent is willing to pay an additional $1.60 for the sugary drink compared to the non-sugary alternative.
Time Frame: 1 week after recruitment (during Part II of the experiment)
Measure: Mean (Standard Deviation); unit: Dollars per 12-pack of soda
Arm/Group | Control Arm | Graphic Warning Labels Arm | Nutrition Labels Arm | Text Warning Labels Arm
Number analyzed (Participants) | 129 | 120 | 115 | 107
Dollars per 12-pack of soda | 0.02 (0.69) | -0.31 (1.02) | -0.58 (1.22) | -0.23 (1.02)
Statistical Analysis 1: Comparison: Control Arm vs Graphic Warning Labels Arm; Test type: Superiority; p = 0.003, Regression, Linear; Treatment Effect = -0.33, 95% CI 2-sided [-0.55 to -0.11]
Statistical Analysis 2: Comparison: Control Arm vs Nutrition Labels Arm; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.61, 95% CI 2-sided [-0.87 to -0.35]
Statistical Analysis 3: Comparison: Control Arm vs Text Warning Labels Arm; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.25, 95% CI 2-sided [-0.48 to -0.17]

3. Other Pre Specified Outcome: Willingness to Purchase Sugar-sweetened Beverage vs. Sugar-free Alternative, by Subgroups
Description: How much different groups of consumers like, or are willing to pay for, sugar-sweetened beverages when compared to a sugar-free alternative. The survey instrument uses a multiple price list (MPL) to elicit each respondent's relative willingness to pay (WTP) for the sugary drink vs. the non-sugary alternative, a standard methodology in the economics literature where consumers answer a series of questions about whether they would prefer to buy a sugar-sweetened beverage at price X or a sugar-free alternative at price Y. For example, a relative WTP of $1.60 indicates a respondent is willing to pay an additional $1.60 for the sugary drink compared to the non-sugary alternative.
Time Frame: 1 week after recruitment (during Part II of the experiment)
Population: We report on gender, race, and ethnicity subgroups. Because each row represents one such subgroup, the number analyzed is by definition smaller than the overall number analyzed. For example, there are 667 participants in the Control Arm, but only 316 of these identified as Male.
Measure: Mean (Standard Deviation); unit: Dollars per 12-pack of soda
Arm/Group | Control Arm | Graphic Warning Labels Arm | Nutrition Labels Arm | Text Warning Labels Arm
Number analyzed (Participants) | 667 | 653 | 644 | 662
Dollars per 12-pack of soda
  Gender: Female or other: number analyzed (Participants) | 351 | 339 | 340 | 364
  Gender: Female or other | 0.03 (0.90) | -0.47 (1.38) | -0.39 (1.20) | -0.26 (1.00)
  Gender: Male: number analyzed (Participants) | 316 | 314 | 304 | 298
  Gender: Male | 0.09 (0.77) | -0.45 (1.30) | -0.40 (1.26) | -0.33 (1.07)
  Race: American Indian or Alaska Native: number analyzed (Participants) | 9 | 6 | 5 | 5
  Race: American Indian or Alaska Native | 0.38 (1.38) | -1.56 (2.23) | -0.05 (0.21) | 0.02 (0.39)
  Race: Asian: number analyzed (Participants) | 34 | 37 | 37 | 40
  Race: Asian | -0.03 (0.88) | -0.71 (1.46) | -0.59 (1.33) | -0.56 (1.30)
  Race: Native Hawaiian or Pacific Islander: number analyzed (Participants) | 1 | 1 | 2 | 1
  Race: Native Hawaiian or Pacific Islander | -0.80 (0.80) | 0.00 (0.00) | -0.80 (0.69) | 0.00 (0.00)
  Race: Black or African American: number analyzed (Participants) | 17 | 29 | 24 | 25
  Race: Black or African American | -0.57 (1.46) | -0.13 (1.83) | -0.32 (1.34) | -0.61 (1.63)
  Race: White: number analyzed (Participants) | 563 | 551 | 548 | 551
  Race: White | 0.07 (1.19) | -0.44 (1.66) | -0.37 (1.65) | -0.26 (1.35)
  Race: More Than One Race: number analyzed (Participants) | 26 | 18 | 14 | 19
  Race: More Than One Race | 0.18 (0.90) | -0.77 (1.89) | -0.99 (2.12) | -0.22 (0.94)
  Race: Unknown or Not Reported: number analyzed (Participants) | 17 | 11 | 14 | 21
  Race: Unknown or Not Reported | 0.12 (0.88) | -0.39 (1.54) | -0.23 (1.22) | -0.17 (1.57)
  Ethnicity: Hispanic: number analyzed (Participants) | 28 | 26 | 27 | 48
  Ethnicity: Hispanic | -0.13 (0.72) | 0.09 (1.50) | -0.31 (1.17) | -0.12 (1.05)
  Ethnicity: Not Hispanic: number analyzed (Participants) | 601 | 592 | 584 | 595
  Ethnicity: Not Hispanic | 0.05 (0.83) | -0.48 (1.34) | -0.40 (1.23) | -0.31 (1.03)
  Ethnicity: Other / Prefer Not To Say: number analyzed (Participants) | 38 | 35 | 33 | 19
  Ethnicity: Other / Prefer Not To Say | 0.36 (1.03) | -0.55 (1.17) | -0.42 (1.32) | -0.2 (1.16)
Statistical Analysis 1: Comparison: Control Arm vs Graphic Warning Labels Arm; Gender subgroup: Female or other; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.5, 95% CI 2-sided [-0.67 to -0.32] — Unit: $ per 12-pack
Statistical Analysis 2: Comparison: Control Arm vs Graphic Warning Labels Arm; Gender subgroup: Male; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.53, 95% CI 2-sided [-0.70 to -0.36] — Unit: $ per 12-pack
Statistical Analysis 3: Comparison: Control Arm vs Nutrition Labels Arm; Gender subgroup: Female or other; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.41, 95% CI 2-sided [-0.57 to -0.25] — Unit: $ per 12-pack
Statistical Analysis 4: Comparison: Control Arm vs Nutrition Labels Arm; Gender subgroup: Male; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.48, 95% CI 2-sided [-0.65 to -0.32] — Unit: $ per 12-pack
Statistical Analysis 5: Comparison: Control Arm vs Text Warning Labels Arm; Gender subgroup: Female or other; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.28, 95% CI 2-sided [-0.42 to -0.14] — Unit: $ per 12-pack
Statistical Analysis 6: Comparison: Control Arm vs Text Warning Labels Arm; Gender subgroup: Male; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.57, 95% CI 2-sided [-0.57 to -0.27]; Unit: $ per 12-pack
Statistical Analysis 7: Comparison: Control Arm vs Graphic Warning Labels Arm; Race subgroup: American Indian or Alaska Native; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -2.23, 95% CI 2-sided [-3.34 to -1.12] — Unit: $ per 12-pack
Statistical Analysis 8: Comparison: Control Arm vs Graphic Warning Labels Arm; Race subgroup: Asian; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.69, 95% CI 2-sided [-1.15 to -0.23] — Unit: $ per 12-pack
Statistical Analysis 9: Comparison: Control Arm vs Graphic Warning Labels Arm; Race subgroup: Native Hawaiian or Pacific Islander; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = 0.80, 95% CI 2-sided [0.80 to 0.80] — Unit: $ per 12-pack
Statistical Analysis 10: Comparison: Control Arm vs Graphic Warning Labels Arm; Race subgroup: Black or African American; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = 0.45, 95% CI 2-sided [-0.24 to 1.14] — Unit: $ per 12-pack
Statistical Analysis 11: Comparison: Control Arm vs Graphic Warning Labels Arm; Race subgroup: White; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.50, 95% CI 2-sided [-0.63 to -0.37] — Unit: $ per 12-pack
Statistical Analysis 12: Comparison: Control Arm vs Graphic Warning Labels Arm; Race subgroup: More Than One Race; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.96, 95% CI 2-sided [-1.67 to -0.25] — Unit: $ per 12-pack
Statistical Analysis 13: Comparison: Control Arm vs Graphic Warning Labels Arm; Race subgroup: Unknown or Not Reported; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.38, 95% CI 2-sided [-1.16 to 0.40] — Unit: $ per 12-pack
Statistical Analysis 14: Comparison: Control Arm vs Nutrition Labels Arm; Race subgroup: American Indian or Alaska Native; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.44, 95% CI 2-sided [-1.07 to 0.19] — Unit: $ per 12-pack
Statistical Analysis 15: Comparison: Control Arm vs Nutrition Labels Arm; Race subgroup: Asian; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.54, 95% CI 2-sided [-0.91 to -0.17] — Unit: $ per 12-pack
Statistical Analysis 16: Comparison: Control Arm vs Nutrition Labels Arm; Race subgroup: Native Hawaiian or Pacific Islander; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unit: $ per 12-pack
Statistical Analysis 17: Comparison: Control Arm vs Nutrition Labels Arm; Race subgroup: Black or African American; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = 0.16, 95% CI 2-sided [-0.36 to 0.68] — Unit: $ per 12-pack
Statistical Analysis 18: Comparison: Control Arm vs Nutrition Labels Arm; Race subgroup: white; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.44, 95% CI 2-sided [-0.57 to -0.31] — Unit: $ per 12-pack
Statistical Analysis 19: Comparison: Control Arm vs Nutrition Labels Arm; Race subgroup: More Than One Race; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -1.18, 95% CI 2-sided [-2.04 to -0.32] — Unit: $ per 12-pack
Statistical Analysis 20: Comparison: Control Arm vs Nutrition Labels Arm; Race subgroup: Unknown or Not Reported; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.38, 95% CI 2-sided [-0.90 to 0.14] — Unit: $ per 12-pack
Statistical Analysis 21: Comparison: Control Arm vs Text Warning Labels Arm; Race subgroup: American Indian or Alaska Native; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.79, 95% CI 2-sided [-1.54 to -0.04] — Unit: $ per 12-pack
Statistical Analysis 22: Comparison: Control Arm vs Text Warning Labels Arm; Race subgroup: Asian; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.51, 95% CI 2-sided [-0.90 to -0.12] — Unit: $ per 12-pack
Statistical Analysis 23: Comparison: Control Arm vs Text Warning Labels Arm; Race subgroup: Native Hawaiian or Pacific Islander; Test type: Superiority; p < 0.001, Regression, Logistic; Treatment Effect = 0.80, 95% CI 2-sided [0.80 to 0.80] — Unit: $ per 12-pack
Statistical Analysis 24: Comparison: Control Arm vs Text Warning Labels Arm; Race subgroup: Black or African American; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.04, 95% CI 2-sided [-0.79 to 0.71] — Unit: $ per 12-pack
Statistical Analysis 25: Comparison: Control Arm vs Text Warning Labels Arm; Race subgroup: White; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.33, 95% CI 2-sided [-0.44 to -0.22] — Unit: $ per 12-pack
Statistical Analysis 26: Comparison: Control Arm vs Text Warning Labels Arm; Race subgroup: More Than One Race; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.41, 95% CI 2-sided [-0.76 to -0.06] — Unit: $ per 12-pack
Statistical Analysis 27: Comparison: Control Arm vs Text Warning Labels Arm; Race subgroup: Unknown or Not Reported; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.27, 95% CI 2-sided [-0.85 to 0.31] — Unit: $ per 12-pack
Statistical Analysis 28: Comparison: Control Arm vs Graphic Warning Labels Arm; Ethnicity subgroup: Hispanic; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = 0.23, 95% CI 2-sided [-0.45 to 0.91] — Unit: $ per 12-pack
Statistical Analysis 29: Comparison: Control Arm vs Graphic Warning Labels Arm; Ethnicity subgroup: Not Hispanic; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.52, 95% CI 2-sided [-0.65 to -0.39] — Unit: $ per 12-pack
Statistical Analysis 30: Comparison: Control Arm vs Graphic Warning Labels Arm; Ethnicity subgroup: Other or Prefer Not to Say; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.93, 95% CI 2-sided [-1.48 to -0.38] — Unit: $ per 12-pack
Statistical Analysis 31: Comparison: Control Arm vs Nutrition Labels Arm; Ethnicity subgroup: Hispanic; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.16, 95% CI 2-sided [-0.70 to 0.38] — Unit: $ per 12-pack
Statistical Analysis 32: Comparison: Control Arm vs Nutrition Labels Arm; Ethnicity subgroup: Not Hispanic; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.45, 95% CI 2-sided [-0.57 to -0.33] — Unit: $ per 12-pack
Statistical Analysis 33: Comparison: Control Arm vs Nutrition Labels Arm; Ethnicity subgroup: Other or Prefer Not to Say; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.79, 95% CI 2-sided [-1.42 to -0.16] — Unit: $ per 12-pack
Statistical Analysis 34: Comparison: Control Arm vs Text Warning Labels Arm; Ethnicity subgroup: Hispanic; Test type: Superiority; p = 0.980, Regression, Linear; Treatment Effect = 0.01, 95% CI 2-sided [-0.40 to 0.41] — Unit: $ per 12-pack
Statistical Analysis 35: Comparison: Control Arm vs Text Warning Labels Arm; Ethnicity subgroup: Not Hispanic; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.36, 95% CI 2-sided [-0.47 to -0.25] — Unit: $ per 12-pack
Statistical Analysis 36: Comparison: Control Arm vs Text Warning Labels Arm; Ethnicity Subgroup: Other or Prefer Not to Say; Test type: Superiority; p < 0.001, Regression, Linear; Treatment Effect = -0.39, 95% CI 2-sided [-1.03 to 0.25] — Unit: $ per 12-pack

ADVERSE EVENTS:
Time Frame: From enrollment of first participant (October 18, 2021) to completion of final participant (December 22, 2021), roughly 2 months
Groups:
- Stage 1 - Non-Randomized: Subjects did not reach Part II of the experiment, and therefore did not reach the point of randomization. This includes subjects who completed Part I but never started Part II and subjects who started Part I but never finished it.
- Stage 2 - Non-Randomized: Subjects began Part II of the experiment, but did not reach the point of randomization.
Arm/Group | Stage 1 - Non-Randomized | Control Arm | Graphic Warning Labels Arm | Nutrition Labels Arm | Text Warning Labels Arm | Stage 2 - Non-Randomized
All-Cause Mortality (participants affected / at risk) | 0/1203 | 0/696 | 0/683 | 0/668 | 0/683 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/1203 | 0/696 | 0/683 | 0/668 | 0/683 | 0/100
Other Adverse Events (participants affected / at risk) | 0/1203 | 0/696 | 0/683 | 0/668 | 0/683 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05038163/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05038163/SAP_001.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05038163/ICF_002.pdf